CLINICAL TRIAL: NCT02526784
Title: A Multi-Centre, Open-Label, Randomised Trial Evaluating Two Subcutaneous Injection Techniques and Intramuscular Administration of Degarelix in Patients With Prostate Cancer
Brief Title: A Trial Evaluating Two Subcutaneous Injection Techniques and Intramuscular Administration of Degarelix in Patients With Prostate Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 000184; 2015-000357-20 (EudraCT Number)
Record Dates: First submitted 2015-08-17; First posted 2015-08-18 (Estimated); Last update posted 2017-07-05 (Actual); Status verified 2017-07

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Injection A (Active Comparator): Degarelix s.c. standard injections
  Interventions: Drug: degarelix
- Injection B (Experimental): Degarelix s.c. optimised injections
  Interventions: Drug: degarelix
- Injection C (Experimental): Degarelix i.m. injections
  Interventions: Drug: degarelix

INTERVENTIONS:
Drug: degarelix
  Other Names: Firmagon

SUMMARY:
The purpose of this trial is to compare the severity of ISRs (Injection Site Reactions) following degarelix subcutaneous (s.c.) administrations with two different injection techniques and intramuscular (i.m.) administration in patients with hormone dependent prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years with a diagnosis of adenocarcinoma of the prostate (Gleason graded, all stages) where endocrine treatment is indicated.
* Caucasian origin.
* Able to provide written Informed Consent and willing and able to comply with trial procedures.
* Body mass index (BMI) between 18.5-30 kg/m2.
* Has a life expectancy of at least one year.

Exclusion Criteria:

* Current hormonal management of prostate cancer.
* Previous endocrine therapy for prostate cancer within 3 months prior to the screening visit.
* Any medical injection therapy that might interfere with degarelix injections.
* Patients with advanced muscle atrophy or cachexia which in the Investigator's opinion would preclude or pose risks of complications following ventrogluteal i.m. injection of degarelix.
* Any medical condition that could be aggravated or may cause extreme discomfort during the trial period or could cause a moderate risk to a patient (significant heart, renal or liver disease).
* Chronic pain syndrome or any continuous pain reported by the patient that, according to the judgement of the Investigator, could limit the evaluation of injection related pain.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2015-12; Primary Completion 2017-05 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Difference in the average patient reported injection site pain score between patients receiving the optimised and standard s.c. injections, as well as between patients receiving the i.m. and standard s.c. injections | From baseline to month 6
  Assessed by a 10-graded numeric pain rating scale (0=no pain, 10=worst possible pain)

SECONDARY OUTCOMES:
Patient reported injection site pain scores after degarelix starting dose | From starting dose to 6 days after starting dose
  Assessed by a 10-graded numeric pain rating scale (0=no pain, 10=worst possible pain)
Patient reported injection site pain scores after degarelix maintenance doses | From first maintenance dose (month 1) to 6 days after last maintenance dose (month 6)
  Assessed by a 10-graded numeric pain rating scale (0=no pain, 10=worst possible pain)
Difference in skin colour values between pre- and post-injection | From baseline to month 6
  Average of 4 measurements on skin redness at the injection site using DSM II ColorMeter

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (3):
- Tampereen yliopistollinen sairaala (there may be other sites in this country), Tampere, Finland
- Groupe Hospitalier Pellegrin Tripode (there may be other sites in this country), Bordeaux, France
- Universitaetsklinikum Freiburg (there may be other sites in this country), Freiburg im Breisgau, Germany